CLINICAL TRIAL: NCT01001988
Title: Long-term Follow-up of Immunogenicity of a Single Dose of JE-CV in Toddlers in Thailand and the Philippines
Brief Title: Long-term Follow-up of Immunogenicity of a Single Dose of Japanese Encephalitis Chimeric Virus Vaccine (JE-CV) in Toddlers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: JEC05; U1111-1112-2127 (Other: WHO)
Record Dates: First submitted 2009-10-23; First posted 2009-10-27 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Encephalitis; Japanese Encephalitis
Keywords: Encephalitis; Japanese Encephalitis; Japanese Encephalitis Chimeric Virus Vaccine; Toddlers
MeSH Terms: conditions — Encephalitis; Encephalitis, Japanese | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study group (Experimental): Participants received a single dose of JE-CV administered in Study JEC02. In Study JEC05 there were yearly visits with blood samples taken for immunogenicity assessment.
  Interventions: Other: Blood sample; Biological: JE-CV administered in Study JEC02

INTERVENTIONS:
Other: Blood sample — Blood sample for immunogenicity assessment
Biological: JE-CV administered in Study JEC02 — Participants received a single dose of JE-CV at 12 to 18 months of age in Study JEC02. No vaccination was administered in Study JEC05

SUMMARY:
This is a long-term follow-up of the persistence of immune response in participants who previously received a single dose of JE-CV at age 12 to 18 months in Study JEC02 (NCT00735644) . No vaccination was administered during the present long-term follow-up study.

Primary Objective:

* To describe the yearly persistence of humoral immune response to Japanese encephalitis after a single dose of JE-CV

DETAILED DESCRIPTION:
Persistence of immune response will be determined in participants who previously received a single dose of JE-CV at age 12 to 18 months in Study JEC02 (NCT00735644). No vaccination will be given in this study.

ELIGIBILITY:
Inclusion Criteria :

* Provision of Informed Consent Form signed by at least one parent or other legally acceptable representative, and by at least one independent witness if required by local regulations.
* Participant who was vaccinated with JE-CV in JEC02 trial and had a pre-vaccination blood sample at baseline in JEC02 trial.
* Participant and parent/legally acceptable representative able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria :

* Receipt of any JE vaccine other than JE-CV during JEC02 trial and during the period up to inclusion in JEC05 trial.
* Planned participation in another clinical trial up to the first year of the follow-up in the present trial.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 596 (Actual)
Dates: Start 2009-08-07 (Actual); Primary Completion 2013-10-16 (Actual); Study Completion 2013-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (3):
- City of Muntinlupa, Philippines
- Thailand (2):
  - Bangkok
  - Khon Kaen

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled at 3 sites in Thailand and 2 sites in the Philippines.
Pre-assignment Details: A total of 596 participants received a single dose of JE-CV in JEC02 and came to Visit 1 (Year 1) in JEC05; 585 participants were included in the Per Protocol Analysis set.
Groups:
- Study Group: Participants received a single dose of JE-CV in Study JEC02 (NCT00735644)
Period: Overall Study
Arm/Group | Study Group
Started | 596
Completed | 479
Not Completed | 117
Not completed — Protocol Violation | 84
Not completed — Withdrawal by Subject | 18
Not completed — Lost to Follow-up | 15

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all participants in the Per Protocol Analysis Set at Year 1 of JEC05
Groups:
- Study Group: Participants received a single dose of JE-CV in Study JEC02
Arm/Group | Study Group
Number analyzed (Participants) | 585
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 585
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 26.2 (1.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 272
  Male | 313
Region of Enrollment [Number; unit: participants]
  Philippines | 229
  Thailand | 356

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Japanese Encephalitis Seroprotection Following a Single Dose of JE-CV
Description: Seroprotection was defined as the proportion of participants with Japanese encephalitis virus neutralizing antibody titers ≥10 1/dil as measured by a JE 50% plaque reduction neutralization test (PRNT50).
Time Frame: Day 0 (pre-vaccination) from study JEC02, Day 28 post-vaccination from study JEC02, and at Years 1, 2, 3, 4, and 5 post-vaccination
Population: Seroprotection was analyzed in the Per Protocol Analysis Set.
Measure: Number; unit: Percentage of participants
Groups:
- Study Group: Participants received a single dose of Japanese encephalitis chimeric virus vaccine (JE-CV) in Study JEC02 (NCT00735644)
Arm/Group | Study Group
Number analyzed (Participants) | 585
Percentage of participants
  Day 0 (pre-vaccination): number analyzed (Participants) | 583
  Day 0 (pre-vaccination) | 2.6
  Day 28 post-vaccination: number analyzed (Participants) | 574
  Day 28 post-vaccination | 100.0
  Year 1 post-vaccination: number analyzed (Participants) | 584
  Year 1 post-vaccination | 88.2
  Year 2 post-vaccination: number analyzed (Participants) | 541
  Year 2 post-vaccination | 90.0
  Year 3 post-vaccination: number analyzed (Participants) | 505
  Year 3 post-vaccination | 93.1
  Year 4 post-vaccination: number analyzed (Participants) | 484
  Year 4 post-vaccination | 87.6
  Year 5 post-vaccination: number analyzed (Participants) | 478
  Year 5 post-vaccination | 85.4

2. Primary Outcome: Summary of Geometric Mean Titers of Japanese Encephalitis Virus Antibodies Following a Single Dose of a JE-CV
Description: Geometric mean titers of Japanese encephalitis virus antibodies were assessed using the PRNT50 test.
Time Frame: Day 0 (pre-vaccination) from JEC02, Day 28 post-vaccination from JEC02, and at Years 1, 2, 3, 4, and 5 post-vaccination
Population: Geometric mean titers were assessed in the Per Protocol Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | Study Group
Number analyzed (Participants) | 585
Titers (1/dil)
  Day 0 (pre-vaccination): number analyzed (Participants) | 583
  Day 0 (pre-vaccination) | 5.13 [5.06 to 5.21]
  Day 28 post-vaccination: number analyzed (Participants) | 574
  Day 28 post-vaccination | 252 [224 to 284]
  Year 1 post-vaccination: number analyzed (Participants) | 584
  Year 1 post-vaccination | 76.8 [67.4 to 87.6]
  Year 2 post-vaccination: number analyzed (Participants) | 541
  Year 2 post-vaccination | 81.4 [71.7 to 92.6]
  Year 3 post-vaccination: number analyzed (Participants) | 505
  Year 3 post-vaccination | 132 [114 to 153]
  Year 4 post-vaccination: number analyzed (Participants) | 484
  Year 4 post-vaccination | 85.8 [74.7 to 98.6]
  Year 5 post-vaccination: number analyzed (Participants) | 478
  Year 5 post-vaccination | 63.3 [54.8 to 73.0]

ADVERSE EVENTS:
Time Frame: Safety data were not collected in this trial as no vaccine was administered. Only serious adverse events (SAEs) related to the vaccination in study JEC02 were collected. Overall, no related SAEs (including death) were reported from 6 months to 5 years post-vaccination in JEC02.
Arm/Group | Study Group
All-Cause Mortality (participants affected / at risk) | 0/591
Serious Adverse Events (participants affected / at risk) | 0/591
Other Adverse Events (participants affected / at risk) | 0/591

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No